CLINICAL TRIAL: NCT06222567
Title: Assessing the Effect of Additional 5 Minutes Pumping on Expression Volume in Breastfeeding Human Initiating Breastfeeding.
Brief Title: Assessing the Effect of an Additional 5 Minutes Pumping on Milk Output in the First Days After Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OLVG040; WO 22.168 (Other: OLVG)
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pumping individual (Experimental): Clinical indication for pumping
  Interventions: Device: 15 minutes pumping with INITIATE program; Device: 5 minutes extra pumping with MAINTAIN program

INTERVENTIONS:
Device: 15 minutes pumping with INITIATE program — 15 minutes pumping with INITIATE program
Device: 5 minutes extra pumping with MAINTAIN program — Additional 5 minutes extra pumping with MAINTAIN program

SUMMARY:
The study hypothesizes that human who are both breastfeeding and pumping in the first days postpartum have more expression volume with an additional 5 minutes of pumping with Maintain program after pumping with the INITIATE program.

DETAILED DESCRIPTION:
This study aims to assess if expression milk volume could be improved for patients pumping milk for a clinical indication by implementing five minutes more pumping with the MAINTAIN program, a different sucking pattern, to initiate and benefit milk production. The results of this study will provide important information that validates the proposed changes as well as build clear recommendation for using the Symphony program cards in this population.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years old
* Infant was born maximum 4 (96 hours) days ago
* Subject has an clinical indication to pump for reasons
* The subject signs the informed consent documentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Total expression volume in milliliter | T1= 15 minutes, T2=20 minutes
  Expressed milk volume in milliliters between 15 and 20 minutes of pumping

SECONDARY OUTCOMES:
Total expression volume in milliliters according to postpartum inclusion day (day 1,2,3 or 4) and patient characteristic. Milk yielded in milliliters per minute after 15 and 20 minutes pumping. | T1= 15 minutes, T2=20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Fedde Scheele, Prof. Dr., Principal Investigator — OLVG Hospital
Locations (1):
- OLVG Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual data is not shared